CLINICAL TRIAL: NCT02117765
Title: Phase I/II Study of Ustekinumab in Patients With New-onset Type 1 Diabetes
Brief Title: Pilot Clinical Trial of Ustekinumab in Patients With New-onset T1D
Acronym: UST1D
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H14-00939
Record Dates: First submitted 2014-04-07; First posted 2014-04-21 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Type 1 Diabetes
Keywords: T1D; ustekinumab; new-onset; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Four cohorts of 5 subjects will be recruited:
  Group 1: Five subjects will be given Ustekinumab 45mg SC at 0, 4, 16, 28 and 40 weeks.
  Group 2: Five subjects will be given Ustekinumab 90mg SC at 0, 4, 16, 28 and 40 weeks.
  Group 3: Five subjects will be given Ustekinumab 45 mg SC at 0,4 and 16 weeks.
  Group 4: Five subjects will be given Ustekinumab 90mg SC at 0, 4 and 16 weeks.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab
  Other Names: Stelara

SUMMARY:
In type 1 diabetes (T1D), immune defense cells in the body attack and destroy insulin-producing beta cells leaving affected people with a lifelong need for daily insulin injections. Even with insulin injections, blood glucose (sugar) control is imperfect and leads to many health complications and a shortened life span. This is a pilot clinical trial to test the safety of a drug, ustekinumab, in 20 adult subjects with recent-onset T1D. Ustekinumab is currently licensed for use in psoriasis where it has proven to be both highly effective and safe and so the investigators hope to see a similar effect in T1D. This trial will also be used to determine the best dosage and frequency of the drug to be given to people with T1D to help design future studies on the drug's effectiveness. The investigators hope that if the drug can block immune cells soon after the development of diabetes, any remaining insulin-producing cells may be protected, and regenerate, thus producing more insulin so that individuals may be insulin free, or require less insulin.

DETAILED DESCRIPTION:
The investigators will perform an open-label pilot safety study (Phase I/II clinical trial) with a total of 20 adult (18-35 years old) subjects with recent-onset T1D. There will be four study cohorts, which will be recruited sequentially all to the treatment arm: five subjects will be given ustekinumab, 45mg subcutaneously (SC) at 0, 4, 16, 28 and 40weeks, five subjects will be given ustekinumab, 90mg SC at weeks 0, 4, 16, 28 and 40, five subjects will be given 45mg SC at weeks 0, 4 and 16 and five subjects will be given 90mg subcutaneously (SC) at weeks 0, 4 and 16. Recruitment and screening for the pilot study will be completed within the first 6 months. The follow up period is 1 year from the first dose.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of type 1 diabetes mellitus in accordance with the canadian diabetes association criteria.
2. An interval of ≤100 days between the diagnosis and the first dose of the study drug
3. Ability to provide documented informed consent.
4. Male or female, aged 18-35 years inclusive, at the time of the anticipated first dose of the study drug.
5. Evidence of residual functioning β cells. This will be assessed by a C-peptide level over 0.2nmol/L in the MMTT test.
6. Positive for at least one diabetes-related autoantibody.
7. Willing to record all insulin taken and blood glucose levels that are required for monitoring during the study, including reporting any hypoglycaemic events.

Exclusion Criteria:

1. No condition that, in the investigators' judgment, is likely to cause the subject to not be able to understand information in order to provide informed consent.
2. History of malignancy.
3. No significant and/or active disease in any body system that is likely to increase the risk to the subject or interfere with the subject's participation in the study.
4. No significant systemic infection during the 6 weeks before the first dose of the study drug.
5. No history of current or past active tuberculosis infection and no latent tuberculosis.
6. Have used any other investigational drug within the 3 months prior to the first dose and/or intend on using any investigational drug for the duration of the study.
7. Prior or current treatment that is known to cause a significant, ongoing change in the course of T1D or immunological status.
8. Current or prior (within 30 days prior to first study drug dose) use of medications known to influence glucose tolerance.
9. No significant abnormal laboratory values during the screening period, other than those due to T1D.
10. Not pregnant, breastfeeding or planning to become pregnant during the 60 days after the last dose of the study drug.
11. Have not received any live vaccines within 30 days prior to the first study drug dose and are not expected to need to receive a vaccine during the study.
12. No prior allergic reaction, including anaphylaxis, to any component of the study drug product.
13. No prior allergic reaction, including anaphylaxis, to any human, humanized, chimeric or rodent antibody treatment.
14. Have not undergone any major surgery within the 30 day period prior to the first drug dose and not anticipating requiring surgery during the study period.
15. Negative results for Hepatitis B surface antigen and for antibodies to Hepatitis B core antigen, or evidence of Hepatitis B surface antibody > 10 IU, and negative for Hepatitis C. Negative results for HIV and not considered by the investigator to be at high risk for HIV infection.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoints (composite outcome measure) | 12 months
  1. Rate, frequency and severity of all adverse events including; hypoglycemic episodes; injection reactions; hypersensitivity reactions; evidence of infection and posterior leukoencephalopathy syndrome.
  2. Vital signs, standard hematology and chemistry tests, physical examinations.

SECONDARY OUTCOMES:
Immunological Endpoints (composite outcome measure) | 12 months
  1. Immune phenotyping via flow cytometry of all Interleukin (IL)-12, IL-23, IL-17, Interferon(IFN)-γ secreting immune subsets.
  2. Basic immune phenotyping of white blood cell subsets.
  3. Human leukocyte antigen(HLA)- A, B, C, DR, DP, DQ typing.
  4. Fluorospot (ELISpot) analysis for IL-17 and IFN-γ secretion in response to whole insulin and antigens for Cluster of differentiation (CD)8+ and CD4+ T cells .
  5. Luminex assessment of serum cytokines IL-17, IFN-γ, IL-12 and IL-23.
  6. Regulatory T cell : Effector T cell ratio
  7. CD154 based assays to determine diabetogenic antigen specific responses of T helper cells.
  8. Epigenetic assessment of Treg phenotype and function.
Exploratory (composite outcome measure) | 12 months
  1. Mixed-meal tolerance test (MMTT) - stimulated 2-hour C-peptide area under the curve (AUC) at weeks 4, 28 and 52.
  2. Insulin use in units per kg body weight per day at weeks 4, 16, 28, 40 and 52.
  3. HbA1C levels at weeks 4, 16, 28, 40 and 52.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Dutz, MD FRCPC, Principal Investigator — Professor Department of Dermatology and Skin Science University of British Columbia; Ashish Marwaha, BMBCh PhD, Study Director — University of British Columbia; Annika Sun, MSc, Study Director — University of British Columbia
Locations (1):
- BC Diabetes, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Marwaha AK, Chow S, Pesenacker AM, Cook L, Sun A, Long SA, Yang JHM, Ward-Hartstonge KA, Williams E, Domingo-Vila C, Halani K, Harris KM, Tree TIM, Levings MK, Elliott T, Tan R, Dutz JP. A phase 1b open-label dose-finding study of ustekinumab in young adults with type 1 diabetes. Immunother Adv. 2021 Nov 13;2(1):ltab022. doi: 10.1093/immadv/ltab022. eCollection 2022. PMID 35072168
- See also: Website for study centre. — http://www.bcdiabetes.ca/